CLINICAL TRIAL: NCT07027566
Title: Effect of an Experimental Cannabidiol Gel on Tooth Sensitivity Induced by Tooth Bleaching
Brief Title: Effect of an Experimental Cannabidiol Gel on Tooth Sensitivity
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Jesuína Lamartine Nogueira Araújo, Principal Investigator: Clinical Professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PPGOUFPAFO
Record Dates: First submitted 2025-05-14; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Dentin Sensitivity
Keywords: Tooth Bleaching; Cannabidiol; Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — potassium nitrate; Sodium Fluoride; Cannabidiol; Gels

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): The placebo gel (PG) (natrosol 4%) will be applied to the buccal surfaces of the central and lateral incisors, canines and upper and lower premolars, with a microbrush actively, for 10 minutes. Subsequently, all groups will undergo in-office whitening treatment with 35% hydrogen peroxide (Whiteness HP, FGM). Sensitivity assessment will be carried out using a form consisting of a visual analogue scale (VAS), patients will be instructed to record tooth sensitivity daily, during the 21 days of follow-up. To measure color, the VITA Easyshade spectrophotometer (VITA, Germany)) will be used at two times: baseline (Ti) and one week after the 3rd bleaching session (Tf).
  Interventions: Drug: Natrosol 4% Gel
- Control group (Active Comparator): gel with 5% potassium nitrate and 2% sodium fluoride The gel with 5% potassium nitrate and 2% sodium fluoride (NKFG) will be applied to the buccal surfaces of the central and lateral incisors, canines and upper and lower premolars, with a microbrush actively, for 10 minutes. Subsequently, all groups will undergo in-office whitening treatment with 35% hydrogen peroxide (Whiteness HP, FGM). Sensitivity assessment will be carried out using a form consisting of a visual analogue scale (VAS), patients will be instructed to record tooth sensitivity daily, during the 21 days of follow-up. To measure color, the VITA Easyshade spectrophotometer (VITA, Germany) will be used at two
  Interventions: Drug: Potassium nitrate and sodium fluoride
- Experimental group (Experimental): The experimental 2% cannabidiol gel (GCBD) will be applied to the buccal surfaces of the central and lateral incisors, canines and upper and lower premolars, with an active microbrush, for 10 minutes. Subsequently, all groups will undergo in-office whitening treatment with 35% hydrogen peroxide (Whiteness HP, FGM). Sensitivity assessment will be carried out using a form consisting of a visual analogue scale (VAS), patients will be instructed to record tooth sensitivity daily, during the 21 days of followup. To measure color, the VITA Easyshade spectrophotometer (VITA, Germany) will be used at two times: baseline (Ti) and one week after the 3rd bleaching session (Tf).
  Interventions: Drug: Cannabidiol (CBD) Gel

INTERVENTIONS:
Drug: Potassium nitrate and sodium fluoride — Gel with 5% potassium nitrate and 2% sodium fluoride gel of 5% potassium nitrate and 2% sodium fluoride for topical application to teeth before bleaching with hydrogen peroxide
  Other Names: GC
  Arms: Control group
Drug: Cannabidiol (CBD) Gel — Cannabidiol gel for teeth ( 2% cannabidiol oil) before bleaching with hydrogen peroxide
  Other Names: GCBD
  Arms: Experimental group
Drug: Natrosol 4% Gel — placebo gel (natrosol-based gel 4%) for topical application to teeth before bleaching with hydrogen peroxide.
  Other Names: GP
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial will be to evaluate the effect applying an experimental gel based on cannabidiol oil (CBD) on tooth sensitivity induced by tooth bleaching with 35% hydrogen peroxide (HP). Volunteers will be selected and allocated to the following groups: GP - placebo gel, GCBD - experimental cannabidiol gel and GKF - Potassium Nitrate and Sodium Fluoride Gel. In each group, the corresponding desensitizing gel will be applied to on the teeth for 10 minutes. All groups will then undergo in-office whitening treatment with 35% hydrogen peroxide. Patients will be instructed to record tooth sensitivity on a daily basis during the 21 days of follow-up. Pain intensity will be measured using a visual analog scale (VAS), while the risk of developing sensitivity will be recorded after each session of the whitening procedure, with two response option.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at least 28 teeth in the cavity
* Good oral and general health

Exclusion Criteria:

* active caries or periodontal disease
* visible cracks in front teeth upper or lower
* with evident malocclusion
* restorations and prosthetics in teeth anterior teeth
* gastroesophageal disorders
* severe internal tooth discoloration (tetracycline , fluorosis or pulped teeth)
* dentin exposure in anterior teeth and /or later
* parafunctional habits
* tooth sensitivity
* whitening treatment prior to or undergoing orthodontic treatment
* Furthermore, smokers, pregnant or breastfeeding women do not will be included.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Measure Degree of Tooth Sensitivity (pain) by a visual analog scale (VAS) After Tooth Whitening | immediately after the intervention, and for a period of 21 days of treatment
  Experimental cannabidiol and gel (experimental group) and potassium nitrate gel (control group) can change sensitivity related to tooth whitening with hydrogen peroxide 35%. So it is necessary measure this pain. The volunteers will mark on the scale (VAS) the level (1-10) of sensitivity immediately after the intervention, and for a period of 21 days of treatment.

SECONDARY OUTCOMES:
Change in Color of Teeth Bleached by spectrophotometer (VITA Easyshade)(quantitative method: (ΔE00) | There will be two colors readings: - 1: Ti: Base line (Until star first bleaching session); - 2: Tf: one week after the last bleaching session.
  Silicone trays will be made, with canine-by-canine impressions. A window will be created on the vestibular surface of each canine of the silicone guide using a metal device with a radius of 6 mm, corresponding to the diameter of the spectrophotometer tip. The tip of the device will be inserted into the silicone guide to obtain the color parameters of the CIEL*a*b* system, where L* represents the value (light or dark); a* is a measurement of red (a* positive) or green (a* negative); b* is a measurement of yellow (b* positive) or blue (b* negative). The sum of the measured values of the upper canines will be used to obtain the averages of each L*a*b* coordinate for each patient. ΔL*, Δa* and Δb* will be calculated by the difference between the time intervals. Subsequently, the color difference between baseline (Ti) and one week after the 3rd bleaching session (Tf) will be calculated using the CIEDE2000 formulas (ΔE00).

CONTACTS AND LOCATIONS:
Overall Officials: Jesuína L Nogueira Araújo, PHD, Principal Investigator — Federal University of Pará
Locations (1):
- Federal University of Pará School of Dentistry, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No
Brazilian legislation (LGPD), 13.709/2018

REFERENCES:
- [Background] Sano IS, de Almeida AS, Xavier GMB, Paes YFO, Silva CM, de Freitas MCC, da Costa RS, Araujo JLN. Synthesis of an experimental gel containing cannabidiol oil and evaluation of effects on bleached bovine enamel. Odontology. 2026 Jan;114(1):108-120. doi: 10.1007/s10266-025-01105-5. Epub 2025 Apr 19. PMID 40253312